CLINICAL TRIAL: NCT03831867
Title: Effectiveness of Pilates on Sagittal Spine Posture, Flexibility, Back Pain, Quality of Life and Anthropometrics Variables on Adolescents: A Randomized Controlled Trial
Brief Title: Changes in Sagittal Spine Posture and Flexibility on Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Noelia González-Gálvez, PhD. Noelia González Gálvez, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGonzalez
Record Dates: First submitted 2019-01-30; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Adolescent Behavior
Keywords: spine; extensibility; children; health; pilates; exercise; physical activity; physical education
MeSH Terms: conditions — Adolescent Behavior; Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): This group is the experimental group. The intervention program consisted on performance Pilates method exercise program during the sessions of Physical Education.
  Interventions: Other: Pilates
- Control (No Intervention): Adolescents assigned to the CG did not receive any structured exercise programme; they just attended their usual Physical Education sessions.

INTERVENTIONS:
Other: Pilates — The intervention program consisted in the realization of exercises of the Pilates Method. The duration of the program was 32 weeks, with a frequency of two weekly sessions and a duration per intervention of 10 minutes. During this time the experimental group developed the intervention program with the Pilates Method.
  Arms: Pilates

SUMMARY:
Several research show a high prevalence of spinal misalignments and a lack of stability of the spine in the adolescent population. In addition, back pain in adolescents is correlated with a longer time spent in sedentary activities, less time of physical activity, higher BMI, body fat percentage and / or the waist-hip index.

Therefore, the main aim of this project were assess the effect of a 10-minute Pilates program carried out in the final part of the Physical Education sessions for 4.5 months and 9 months on back pain, quality of life, sagittal spine curvature, hamstring extensibility, BMI, body fat percentage and the waist-hip index.

The present research will be elaborated by a quasi-experimental design, with experimental group (GE) and control group (CG); with pre-test, intermediate and post-test.

The inclusion criteria will be: a) being in Compulsory Secondary Education; b) not present any musculoskeletal, neurological, cardiological, metabolic, rheumatic or previous history of spinal pathologies or with previous treatment; c) be active in the sessions of Physical Education.

It was assessed back pain with Back Pain Survey in adolescents. Quality of life was assessed through the Kidscreen-27 questionnaire. To assess the sagittal spinal curvatura (in several positions) the Spinal Mouse System (Idiag, Fehraltdorf, Switzerland) was used.

The extensibility of hamstring muscle was assessed with seat and reach test, toe touch test and active and passive straight leg raising test.

The sedentary lifestyle as well as the level of physical activity will be evaluated through the Adolescent International Physical Activity Questionnaire (IPAQ).

The body mass index will be obtained by recording weight and height (BMI = Weight (kg) / height (cm) 2).

The waist-hip ratio is the quotient between waist and hip circumferences, which is an indirect marker of intra-abdominal obesity.

The intervention program consisted on performance of exercises of the Pilates Method during the sessions of Physical Education, 32 weeks, two weekly sessions, 10 minutes.

DETAILED DESCRIPTION:
A history of back pain during adulthood is related to a history of back pain during adolescence. Therefore, preventing back pain in adolescents helps to prevent their appearance in adulthood. Sagittal spinal misalignments and stability of the spine are in connection with back pain in adolescents. In addition, they influence on several spinal pathologies and decrease the functional capacity and quality of life of adolescents.

Therefore, the objectives of the following project were: a) assess back pain in schoolchildren and check their relationship with quality of life, sagittal spine curvature, extensibility of the hamstring muscles, sedentary lifestyle, physical activity, BMI , percentage of body fat and the waist-hip index; b) measure the sagittal spinal curvature of the schoolchildren, the quality of life and the prevalence of physical activity among adolescents and check their relationship with the hamstring extensibility, sedentary lifestyle, the BMI , percentage of body fat and the waist-hip index; c) analyze the effect of a 10-minute Pilates program carried out in the final part of the Physical Education sessions for 4.5 months and 9 months on back pain, quality of life, sagittal spinal curvatures, the hamstring flexibility, the BMI, the percentage of body fat and the waist-hip index.

The present investigation will be elaborated by a quasi-experimental design, with experimental group (GE) and control group (CG); with pre-test, intermediate and post-test, with analysis of intra-group and inter-group measurements for each of the dependent variables selected in the study.

The inclusion criteria will be: a) being in Compulsory Secondary Education; b) not present any musculoskeletal, neurological, cardiological, metabolic, rheumatic or previous history of spinal pathologies or with previous treatment; c) be active in the sessions of Physical Education.

It was assessed back pain with Back Pain Survey in adolescents. Quality of life was assessed through the Kidscreen-27 questionnaire. To assess the sagittal spinal curvatura (in several position) the Spinal Mouse System (Idiag, Fehraltdorf, Switzerland) was used.

The extensibility of hamstring muscle was assessed with seat and reach test, toe touch test and active and passive straight leg raising test.

The sedentary lifestyle as well as the level of physical activity will be evaluated through the Adolescent International Physical Activity Questionnaire (IPAQ).

The body mass index will be obtained by recording weight and height (BMI = Weight (kg) / height (cm) 2).

The waist-hip ratio is the quotient between waist and hip circumferences, which is an indirect marker of intra-abdominal obesity.

The intervention program consisted in the realization of exercises of the Pilates Method during the sessions of Physical Education. The duration of the program will be 32 weeks, with a frequency of two weekly sessions and a duration per intervention of 10 minutes. During this time the experimental group developed the intervention program with the Pilates Method and the control group carried out their usual sessions of Physical Education . All students to be taken into account in the research must have attended and conducted the practice at least 80% of sessions. The program consisted of four Pilates exercises, planned with a basic-intermediate level, gradually incorporating the Principles of the Pilates Method and increasing the intensity of the exercises. Among these four exercises, two focus on the work of the resistance of the flexor muscles of the trunk, one in the work of the resistance of the trunk extensor musculature and another in the work of hamstring extensibility.The exercises will be performed in cool down of the sessions of Physical Education.

ELIGIBILITY:
Inclusion Criteria:

* be enrolled in Compulsory Secondary Education
* be active in the sessions of Physical Education.

Exclusion Criteria:

* presenting any musculoskeletal, neurological, cardiological, metabolic or rheumatic alteration
* missing more than one session of the programme (91.66% attendance)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 286 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change Sagittal spinal curvature | Change from Baseline Sagittal spinal curvature at 4,5 month and at 9 month
  Sagittal spinal curvature is assess with the Spinal Mouse System. It is measure: angle of the dorsal and lumbar curve and pelvic tilt when standing, in self-correcting standing, in asthenic sitting, in maximum trunk flexion. knees flexed and extended; and maximum trunk flexion from standing. This is noninvasive technique. The result is register in grades.
Change Hamstring extensibility - active straight leg raising test. | Change from Baseline hamstring extensibility at 4,5 month and at 9 month
  The hamstring extensibility is assessed by active straight leg raising test. This is noninvasive technique. The result is register in grades. Higher values represent a better outcome. The range could be between 0 to 180º. Normal values: between 75 to 180º; Shortness type I: between 61 to 74º; and shortness type II; less than 60º. Shortness is mean that the subject have less hamstring extensibility than the normal.
Change Hamstring extensibility - passive straight leg raising test. | Change from Baseline Hamstring extensibility at 4,5 month and at 9 month
  The hamstring extensibility is assessed by passive straight leg raising test. This is noninvasive technique. The result is register in grades. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Change Back pain, physical activity and sedentary behaviour (questionnaire) | Change from Baseline Sagittal spinal curvature at 4,5 month and at 9 month
  Back pain, physical activity and sedentary behaviour is evaluated through the Back Pain Survey in adolescents. This questionnaire included questions about this three items.
  This survey is used to know the prevalence of back pain, physical activity and sedentary time.
  The survey do not includes a scale. The survey ask questions like: Did you have back pain last year that will hamper or limit activities at school or in their leisure time for more than 3 months? Yes/no ; Do you practice any sport in your free live? Yes/No
Change Quality of life: Kindscreem 27 questionnaire | Change from Baseline Back pain, physical activity and sedentary behaviour at 4,5 month and at 9 month
  Quality of life is assessed through the Kindscreem 27 questionnaire.
  To measure the quality of life related to health in adolescents with a total of 27 items assessed on the Likert Scale in the following dimensions: physical activity and health, psychological well-being, relationship with peers and autonomy, social support and peers, and the environment school. Categorizing:
  Extremely difficult 27 to 54;Moderate difficulty 55 to 81;No difficulty makes 82 to 135
Change Body mass index | Change from Baseline Body mass index at 4,5 month and at 9 month
  The body mass index is obtained by recording weight and height. They will be measured with a 220k digital medical scale with height meter. The BMI will be calculated with the formula of the Quetelet Index (1869) (BMI = Weight (kg) / height (cm) 2).
Change Waist-hip ratio | Change from Baseline Waist-hip ratio at 4,5 month and at 9 month
  The waist-hip ratio is the quotient between waist and hip circumferences, which is an indirect marker of intra-abdominal obesity. This is noninvasive technique.
Change Hamstring extensibility Seat and Reach test | Change from Baseline Hamstring extensibility at 4,5 month and at 9 month
  The hamstring extensibility is assessed by seat and reach test. This is noninvasive test.
  The result is register in centimeters. Higher values represent a better outcome.
Change Hamstring extensibility Toe touch test | Change from Baseline Hamstring extensibility at 4,5 month and at 9 month
  The hamstring extensibility is assessed by toe touch test. This is noninvasive test.
  The result is register in centimetres. Higher values represent a better outcome.
Change Level of physical activity - Adolescent International Physical Activity Questionnaire (IPAQ). | Change from Baseline Level of physical activity at 4,5 month and at 9 month
  The level of physical activity will be evaluated through the Adolescent International Physical Activity Questionnaire (IPAQ).
  It is register and summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.The following values continue to be used for the analysis of IPAQ data: Walking=3.3METs (equivalent metabolic), Moderate PA (physical activity)=4.0METs (Metabolic equivalent) and Vigorous PA=8.0METs (Metabolic equivalent).
  Category 1 Low: Those individuals who not meet criteria for Categories 2 or 3. Category 2 Moderate: Total physical activity of at least 600 MET-minutes/week. Category 3 High: a) Total physical activity of at least 3000 MET-minutes/week.

CONTACTS AND LOCATIONS:
Overall Officials: Noelia G Gálvez, PhD., Principal Investigator — UCAM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson L, Haladay DE. Pilates-based exercise in the treatment of a patient with persistent low back pain following transforaminal lumbar interbody fusion. Physiother Theory Pract. 2020 Apr;36(4):542-549. doi: 10.1080/09593985.2018.1488905. Epub 2018 Jun 26. PMID 29944036
- [Background] Cruz-Diaz D, Romeu M, Velasco-Gonzalez C, Martinez-Amat A, Hita-Contreras F. The effectiveness of 12 weeks of Pilates intervention on disability, pain and kinesiophobia in patients with chronic low back pain: a randomized controlled trial. Clin Rehabil. 2018 Sep;32(9):1249-1257. doi: 10.1177/0269215518768393. Epub 2018 Apr 13. PMID 29651872
- [Background] Miyamoto GC, Franco KFM, van Dongen JM, Franco YRDS, de Oliveira NTB, Amaral DDV, Branco ANC, da Silva ML, van Tulder MW, Cabral CMN. Different doses of Pilates-based exercise therapy for chronic low back pain: a randomised controlled trial with economic evaluation. Br J Sports Med. 2018 Jul;52(13):859-868. doi: 10.1136/bjsports-2017-098825. Epub 2018 Mar 10. PMID 29525763
- [Background] Kibar S, Yardimci FO, Evcik D, Ay S, Alhan A, Manco M, Ergin ES. Can a pilates exercise program be effective on balance, flexibility and muscle endurance? A randomized controlled trial. J Sports Med Phys Fitness. 2016 Oct;56(10):1139-1146. Epub 2015 Oct 16. PMID 26473443
- [Background] Vaquero-Cristobal R, Lopez-Minarro PA, Alacid Carceles F, Esparza-Ros F. [THE EFFECTS OF THE PILATES METHOD ON HAMSTRING EXTENSIBILITY, PELVIC TILT AND TRUNK FLEXION]. Nutr Hosp. 2015 Nov 1;32(5):1967-86. doi: 10.3305/nh.2015.32.5.9678. Spanish. PMID 26545650
- [Background] Miranda IF, Souza C, Schneider AT, Chagas LC, Loss JF. Comparison of low back mobility and stability exercises from Pilates in non-specific low back pain: A study protocol of a randomized controlled trial. Complement Ther Clin Pract. 2018 May;31:360-368. doi: 10.1016/j.ctcp.2017.12.005. Epub 2017 Dec 8. PMID 29248397
- [Background] Gonzalez-Galvez N, Marcos-Pardo PJ, Carrasco-Poyatos M. Functional improvements after a pilates program in adolescents with a history of back pain: A randomised controlled trial. Complement Ther Clin Pract. 2019 May;35:1-7. doi: 10.1016/j.ctcp.2019.01.006. Epub 2019 Jan 10. PMID 31003644
- [Derived] Gonzalez-Galvez N, Marcos-Pardo PJ, Albaladejo-Saura M, Lopez-Vivancos A, Vaquero-Cristobal R. Effects of a Pilates programme in spinal curvatures and hamstring extensibility in adolescents with thoracic hyperkyphosis: a randomised controlled trial. Postgrad Med J. 2023 Jun 8;99(1171):433-441. doi: 10.1136/postgradmedj-2021-140901. PMID 37294727